CLINICAL TRIAL: NCT05983744
Title: Pulsatile Perfusion Therapy Phase II: A Novel Approach for Improving Cerebral Tissue Blood Flow and Oxygenation
Brief Title: Pulsatile Perfusion Therapy Phase II
Acronym: PPT2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Caroline Rickards (Other)
Responsible Party: Sponsor-Investigator, Caroline Rickards, Associate Professor, University of North Texas Health Science Center
Organization: University of North Texas Health Science Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: IRB #2019-046
Record Dates: First submitted 2021-11-23; First posted 2023-08-09 (Actual); Last update posted 2023-08-09 (Actual); Status verified 2023-08

CONDITIONS: Hemorrhage
MeSH Terms: conditions — Hemorrhage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pulsatile perfusion therapy (PPT) (Experimental): Application of oscillatory lower body negative pressure (LBNP) at specific target frequencies of interest.
  Interventions: Other: 0 Hz Control; Other: 0.1 Hz PPT; Other: 0.05 Hz PPT

INTERVENTIONS:
Other: 0 Hz Control — Lower body negative pressure (LBNP) applied to -60 mmHg for 10-min
Other: 0.1 Hz PPT — Lower body negative pressure (LBNP) applied at a frequency of 0.1 Hz from -30 mmHg to -90 mmHg
Other: 0.05 Hz PPT — Lower body negative pressure (LBNP) applied at a frequency of 0.05 Hz from -30 mmHg to -90 mmHg

SUMMARY:
Individuals who suffer from a stroke, cardiac arrest, or traumatic bleeding (hemorrhage) injuries often have compromised blood flow and oxygen to the brain which can lead to the death of brain cells, and if the patient survives, subsequent difficulty in thinking and performing tasks of daily living. Traditionally, delivery of a constant flow of blood to the brain has been thought to be the most important factor for the survival of brain cells. In this study, a novel intervention will be assessed called "pulsatile perfusion therapy", delivering blood flow in a slow pulsing pattern. It is anticipated this intervention will improve brain blood flow and oxygenation during these serious clinical events.

There is a specific interest in whether delivery of brain blood flow with a slow pulsatile pattern will improve oxygenation of brain tissue, particularly when the brain is challenged under low oxygen (hypoxia) and low volume (hypovolemia) conditions, simulating stroke, cardiac arrest, and hemorrhage. A technique called oscillatory lower body negative pressure (OLBNP) will be used in healthy human participants, facilitating delivery of blood flow to the brain with different pulsing patterns. This technique will allow for determination of the ideal pattern of brain blood flow that improves oxygenation of the brain tissue. Measurements will be made of substances in the blood that may be released with pulsatile flow which act on the blood vessels to increase flow and delivery of oxygen.

DETAILED DESCRIPTION:
Hemorrhage due to trauma is one of the leading causes of morbidity and mortality worldwide in both the civilian and military settings. A major factor contributing to death and disability from severe blood loss is poor tissue perfusion and oxygenation of the vital organs. Traditionally, protection of absolute cerebral blood flow (CBF) has been deemed the most important factor in maintaining perfusion and oxygenation. In recent years, it has been shown that low frequency (LF, ~0.1 Hz) pulsatile CBF is associated with increased tolerance to simulated hemorrhage in healthy human subjects, despite ≥30% reductions in absolute CBF. The underlying mechanism for this improvement in tolerance is unclear; the proposed study aims to address this knowledge gap. The central hypothesis is that LF oscillations (~0.1 Hz) will improve CBF and tissue oxygenation under hypoxic and/or hypovolemic conditions, due to increased shear stress and the release of vasoactive mediators that facilitate vasodilation and enhanced tissue perfusion. This hypothesis will be addressed in two Specific Aims under hypoxic and hypovolemic conditions: 1) determine if inducing oscillations in arterial blood pressure and CBF at 0.1 Hz elicits shear stress-induced vasodilation, subsequently increasing CBF and oxygenation; and, 2) assess the effect of 0.1 Hz oscillations on the release of shear stress-induced vasoactive mediators. Twenty human subjects (males and females) will be recruited to address these aims using oscillatory lower body negative pressure (OLBNP) to induce 0.1 Hz oscillations. Measurements will include CBF (intracranial & extracranial arteries), shear stress, cerebral oxygenation, arterial pressure, and venous blood samples for assessment of nitric oxide, prostaglandin E2, 6-keto-PGF1α (a metabolite of prostacyclin, PGI2), histamine, and endothelin-1. The rationale for the proposed research is to identify a mechanism for the previously observed increase in tolerance to simulated hemorrhage with increases in LF oscillations in arterial pressure and CBF. The approach is innovative as it challenges the traditional association of hemodynamic variability with negative clinical outcomes using a novel methodological approach in human subjects. This contribution is significant as the findings may provide an alternative approach to maintaining cerebral perfusion and oxygenation under conditions of hypovolemia and/or hypoxia.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 to 40 years
2. Non-tobacco/nicotine users (e.g., cigarettes (including electronic cigarettes), chewing tobacco, nicotine gum or patches)
3. Systolic arterial pressure <140 mmHg; diastolic arterial pressure <90 mmHg
4. Normal 12-lead ECG (reviewed by a physician)
5. Normal clinical results from a medical exam reviewed by a board certified physician (e.g., General Health Questionnaire - see attached document)
6. Easily visualized internal carotid and vertebral arteries (via Doppler ultrasound) for accurate measurement of velocity and diameter.
7. Body mass index (BMI) <30 kg/m2 unless athletic/muscular build; calculation = body weight (kg)/height (m2); this criteria is used to ensure subjects will fit inside the LBNP chamber
8. Females only: documentation of a negative pregnancy test prior to the familiarization and experimental sessions

Exclusion Criteria:

1. Age <18 or >40 years
2. Use of tobacco/nicotine within the last 6 months (e.g., cigarettes (including electronic cigarettes), chewing tobacco, nicotine gum or patches)
3. Body mass index (BMI) >30 kg/m2 unless athletic/muscular build; calculation = body weight (kg)/height (m2)
4. Not abstaining from the following 24 hours prior to the experimental session: exercise, alcoholic substances, prescription or non-prescription medications (unless cleared by the medical screener), dietary supplements, herbal medications, caffeinated substances (including coffee, tea (iced or hot), caffeinated energy drinks or sodas).
5. Inability to visualize the internal carotid and vertebral arteries (via Doppler ultrasound) for accurate measurement of velocity and diameter.
6. Positive pregnancy test
7. Post-menopausal females
8. Females with an erratic/irregular menstrual cycle
9. Use of prescription drugs, non-prescription drugs or herbal medicines known to alter cardiovascular, autonomic, or cerebrovascular function unless cleared prior to the study
10. Use of anti-hypertensive medications
11. Use of beta blockers
12. Frequent use of bronchodilators (occasional use, i.e. seasonally, is allowable)
13. Use of anti-coagulant therapy
14. Use of non-contraceptive related hormone therapy
15. Current or past history of hyperthyroidism, or other thyroid hormone-related disease
16. Signs of cardiovascular abnormalities (e.g., resting systolic blood pressure >140mmHg or diastolic blood pressure >90mmHg; abnormal 12-lead ECG)
17. History of cerebrovascular abnormalities (e.g., prior stroke, transient ischemic attacks, epilepsy)
18. Known history of atherosclerosis of the carotid arteries (i.e., plaque formation)
19. History of concussion and or other loss of consciousness within the preceding month
20. Autonomic dysfunction (e.g., Shy-Drager Syndrome, Bradbury-Eggleston syndrome, sinus arrhythmia, idiopathic orthostatic hypotension, fainting disorder)
21. Respiratory illnesses (e.g., chronic asthma (including exercise-induced asthma), Chronic Obstructive Pulmonary Disease, Reactive Airway Disease)
22. History of anaphylaxis
23. Known allergies to medications or other substances (e.g. latex) unless cleared prior to the study
24. History of pre-syncopal/syncopal episodes or orthostatic hypotension
25. Donated blood within the last 60 days
26. History or family history of abnormal blood clotting, clots in deep veins in the legs or pelvis, or blood clots to the lungs aa) Known or suspected abdominal hernia bb) History of alcohol or drug abuse which inhibits the subject's ability to complete this study cc) Known depression, anxiety, or any other mental health issue which inhibits the subject's ability to complete this study dd) Known claustrophobia ee) Previous positive diagnosis of COVID-19

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2020-02-27 (Actual); Primary Completion 2021-12-17 (Actual); Study Completion 2021-12-17 (Actual)

PRIMARY OUTCOMES:
Change in ScO2 | Up to 3-months
  Cerebral tissue oxygen saturation
Change in ICA flow | Up to 3-months
  Internal carotid artery blood flow
Change in MCA velocity | Up to 3-months
  Middle cerebral artery velocity
Change in circulating vasoactive mediators | Up to 3-months
  Venous plasma nitric oxide and endothelin

SECONDARY OUTCOMES:
Change in arterial pressure | Up to 3-months
  Systolic, diastolic, and mean arterial pressure
Change in heart rate | Up to 3-months
  Heart rate
Change in stroke volume | Up to 3-months
  Stroke volume
Change in PCA velocity | Up to 3-months
  Posterior cerebral artery velocity
Change in etO2 and etCO2 | Up to 3-months
  End-tidal oxygen and carbon dioxide

CONTACTS AND LOCATIONS:
Locations (1):
- University of North Texas Health Science Center, Fort Worth, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie the results in a publication
Supporting Information: Study Protocol
Time Frame: Starting 6 months after publication.